CLINICAL TRIAL: NCT01047761
Title: Multi-modal Exercise Program for Chronic Stable Myasthenia Gravis
Brief Title: Exercise for Stable Myasthenia Gravis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Collaborators: University of Maryland (Other)
Responsible Party: Principal Investigator, Charlene Elaine Hafer-Macko, Myasthenia Gravis and Exercise, Baltimore VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Myasthenia and Exercise
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis; Exercise; Fitness; Body Composition; Physical Activity; Pulmonary Function; Balance
MeSH Terms: conditions — Myasthenia Gravis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exercise (Experimental): Multimodal exercises that include walking, breathing exercises, dynamic balance, and core strengthening.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 3 month exercise intervention, three days a week Progressive in duration - up to 1 hour daily; Progressive in intensity
  Multi-modal exercise program includes a) aerobic - walking, b) resistive training with therabands and core exercises, and c) breathing exercises

SUMMARY:
Generalized fatigue in myasthenia gravis results in physical deconditioning that reduces fitness and increases risk of obesity, hypertension, elevated cholesterol and type 2 diabetes. This study will examine how active and fit are 30 individuals with chronic, generalized myasthenic subjects. This study will also determine whether a 3 month home exercise program with aerobic, resistive, and pulmonary training can improve physical activity, strength, fitness, lung function and reduce cardiovascular disease risk.

DETAILED DESCRIPTION:
Generalized fatigue in myasthenia gravis results in a sedentary lifestyle and profound physical deconditioning, leading to reduced fitness and increased risk of obesity, hypertension, dyslipidemia, and type 2 diabetes. This study will characterize the activity and fitness levels and cardiovascular disease risk profile in 30 chronic, generalized myasthenic subjects. Hypotheses are that a) subjects with myasthenia gravis are physically inactive with reduced fitness level and high incidence of obesity and poor cardiovascular disease risk profile, and b) a 3 month multi-modal home exercise program that includes aerobic, resistive, and pulmonary training components will improve physical activity, strength, fitness, dyspnea, body composition and reduce cardiovascular disease risk. Specific aims are to a) define the baseline physical activity and fitness levels and prevalence of insulin resistance and dyslipidemia in stable sedentary myasthenic subjects, b) determine whether a 3 month moderate intensity home exercise program is safe and feasible in deconditioned, stable myasthenic subjects and c) whether a 3 month comprehensive home exercise program can enhance fitness, strength, and lung function to improve physical activity and reduce cardiovascular disease risk.

ELIGIBILITY:
Inclusion Criteria:

* stable generalized myasthenia gravis
* adults age 18-70

Exclusion Criteria:

* already performing regular exercise
* unstable angina
* recent (<3 month) myocardial infarction, stroke, hospitalization for major illness or major surgery
* chronic pain or orthopedic condition restricting exercise
* active cancer, excluding basal cell cancer
* anemia (HCT <30)
* pregnancy
* myasthenia gravis exacerbation in past 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Fitness, Economy of Gait, Physiologic Reserve | Baseline and 3 months

SECONDARY OUTCOMES:
Ambulatory function (6 minute walk, 5 day step activity and accelerometer data) | Baseline and 3 month
Muscle strength by dynamometer | Baseline and 3 month
Myasthenia Quality of Life Scale, SF-36, and Visual Analogue Fatigue Scale | Baseline and 3 months
Cardiovascular risk profile (fasting glucose, oral glucose tolerance test, HbA1c, lipids), smoking status, and body mass index | Baseline and 3 months
Body Composition by DEXA and CT of mid-thigh and hip | Baseline and 3 months
Quantitative MG Scale | Baseline and 3 months
Pulmonary function tests - FVC and maximal inspiratory and expiratory pressure | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Charlene E Hafer-Macko, MD, Principal Investigator — Baltimore VA Medical Center
Locations (1):
- University of Maryland and Baltimore VA Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Myasthenia Gravis Foundation of America — http://www.myasthenia.org/
- See also: University of Maryland Myasthenia Gravis Center — http://www.umm.edu/mg/